CLINICAL TRIAL: NCT05565287
Title: Combining Neonatal Neurobehavioral (Brazelton) And Motor Behavior (Prechtl) In The Assessment And Ultra Early Physical Therapy Intervention Of Premature Infants
Brief Title: Neonatal Neurobehavioral And Motor Behavior In Ultra Early Physical Therapy Intervention
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Moscholouri Chrysoula, Principal Investigator, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MC10107802620
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Disease; Parenting; Premature Birth
Keywords: prematurity; subsystem organization; motor system; state system; general movements; spontaneous mobility; parental confidence; neonatal neurobehavior
MeSH Terms: conditions — Infant, Newborn, Diseases; Premature Birth

STUDY DESIGN:
Intervention Model Description: 1. group: Intervention Parental advise based on the combination of neonatal neurobehaviourism and motor behaviour
  2. group: Basic hospital guidelines
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: prematurity (NICU)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brazelton and Prechtl Assessment Group (Experimental): Parental advise and intervention based on the combination of neonatal neurobehaviourism (Brazelton) and motor behaviour (Prechtl)
  Interventions: Combination Product: ultra early physiotherapy intervention
- No intervention group (No Intervention): Basic hospital guidelines

INTERVENTIONS:
Combination Product: ultra early physiotherapy intervention — * NBAS / NBO and GMs based guidelines in explaining neonatal "signs" into the NICU (lasting 15-30 minutes)
  * NBAS / NBO and GMs based guidelines in explaining neonatal "signs" to parents, 1st neonatal assessment and intervention upon hospital discharge (lasting one hour)
  * NBAS / NBO and GMs based guidelines in explaining neonatal "signs" to parents, 1st neonatal assessment and intervention every 15 to 20 days until the 3rd month of life (corrected age).
  Other Names: Neurobehavioral Concept (Brazelton); Motor Behavioural Concept (Prechtl)
  Arms: Brazelton and Prechtl Assessment Group

SUMMARY:
Investigation of the combination of neonatal neurobehaviourism and motor behavior in the assessment and ultra-early physical therapy intervention of premature neonates and parental support.

DETAILED DESCRIPTION:
Developments in neonatology and perinatal medicine in recent years have resulted in a remarkable development of the survival of premature infants. At the same time, several evaluation and intervention protocols have been developed, aiming at early diagnosis and intervention, but also and studies that are concluding and highlight the need for future well planed and in-depth research, mainly in areas related to early intervention. T. Brazeltons' (1973) Neonatal Behavioural Assessment Scale (NBAS) has been used in many studies of assessment and intervention in newborn-infant and their families and respectively H.R. Prechtls' (1979) Qualitative Assessment of General Movements (GMs) in assessment studies, as a valid and reliable non-invasive procedure. However, the combination of their basic principles and guidelines has not been developed and tested in the context of ultra-early physiotherapy intervention in premature infants.

The evaluation and strengthening of ultra-early physiotherapy intervention by combining basic principles of neonatal neuro-behavior (based on Brazelton T.) and motor behavior (based on Prechtl H.F.R.), in the context of individualized and developmental supportive care of premature neonates and infants and enhancing parental self-confidence.

The research is based upon on three different researches: a) the cross-cultural adaptation of Karitane Parental Confidence Scale (KPCS) questionnaire. The sample will be parents of infants up to one year, b) the effect of ultra-early intervention on parental confidence of preterm infant parents. An experimental randomized controlled trial which will be conducted in the Neonatal Intensive Care Unit (NICU) until maternity hospital discharge. The sample will be premature infants and their parents and c) the effect of ultra-early intervention and parental confidence, on the development of premature infants up to the age of three months. An experimental randomized controlled trial which will be conducted in the Neonatal Intensive Care Unit (NICU) and upon their discharge from the maternity hospital up to the age of 3 months. The study sample will be premature infants and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age under 37 weeks
* Premature newborns hospitalised in the NICU for at least eight days
* (for parents) be able to speak and read Greek or English

Exclusion Criteria:

* Newborns with congenital and chromosomal abnormalities.
* Newborns with severe accompanying pathological problems and congenital infections.
* (for parents) with known history of drug or alcohol abuse or serious psychiatric disorders

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The neonatal behavioural assessment scale (NBAS) | newborn - 2 month old (corrected age)
  Assesses neurobehavioral repertoire of the newborn
The New-born Behavioral Observations (NBO) | Βirth through the 3rd month of life
  latest and inspired by the clinical uses of NBAS. Αn interactive relationship-building tool to strengthen the relationship between infants and parents beginning in the newborn period
The Qualitative Assessment of General Movements (GMsA) | birth to 20 weeks (corrected age)
  non-invasive and non-disruptive assessment through observations of the quality of generalised movements to determine the integrity of the CNS of infants
• Karitane Parenting Confidence Scale (KPCS) (Crncec, R., et all., 2008, 2010) | Birth to 12 months
  Assesses perceived parental confidence in newborn/infant care
• Parental Stressor Scale: Neonatal Intensive Care Unit (Pss: Nicu) (Miles, M. S., Funk, S. G., & Carlson, J., 1993) | From Enrollment to the end of interventional 3 months
  Parental Self Reported Questionnaire concerning their experiences in NICU

SECONDARY OUTCOMES:
Parental Stress Scale (PSS-18) (Berry, J., O., & Jones., W., H., 1995) | From enrollment to the end of program at 3 months
  Parental Self Reported Questionnaire concerning their parental experience

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis N Triggas, Assistant Profesor, Study Director — University of Thessaly
Locations (3):
- Greece (3):
  - PAGNI University Hospital, Heraklion, Crete
  - Attikon Hospital, Athens, Haidari
  - University of Thessaly, Lamia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Als H. The newborn communicates. J Commun. 1977 Spring;27(2):66-73. doi: 10.1111/j.1460-2466.1977.tb01828.x. No abstract available. PMID 853137
- [Background] Aita M, Snider L. The art of developmental care in the NICU: a concept analysis. J Adv Nurs. 2003 Feb;41(3):223-32. doi: 10.1046/j.1365-2648.2003.02526.x. PMID 12581110
- [Background] Volpe JJ. Brain injury in the premature infant--current concepts of pathogenesis and prevention. Biol Neonate. 1992;62(4):231-42. doi: 10.1159/000243876. PMID 1420621
- [Background] Prechtl HF. Qualitative changes of spontaneous movements in fetus and preterm infant are a marker of neurological dysfunction. Early Hum Dev. 1990 Sep;23(3):151-8. doi: 10.1016/0378-3782(90)90011-7. No abstract available. PMID 2253578
- [Background] Bekedam DJ, Visser GH, de Vries JJ, Prechtl HF. Motor behaviour in the growth retarded fetus. Early Hum Dev. 1985 Nov;12(2):155-65. doi: 10.1016/0378-3782(85)90178-1. PMID 3905347
- [Background] Geerdink JJ, Hopkins B. Qualitative changes in general movements and their prognostic value in preterm infants. Eur J Pediatr. 1993 Apr;152(4):362-7. doi: 10.1007/BF01956755. PMID 8482291
- [Background] Craciunoiu O, Holsti L. A Systematic Review of the Predictive Validity of Neurobehavioral Assessments During the Preterm Period. Phys Occup Ther Pediatr. 2017 Aug;37(3):292-307. doi: 10.1080/01942638.2016.1185501. Epub 2016 Jun 17. PMID 27314272
- [Background] Noble Y, Boyd R. Neonatal assessments for the preterm infant up to 4 months corrected age: a systematic review. Dev Med Child Neurol. 2012 Feb;54(2):129-39. doi: 10.1111/j.1469-8749.2010.03903.x. Epub 2011 Dec 5. PMID 22142216
- [Background] Aita M, Stremler R, Feeley N, Lavallee A, De Clifford-Faugere G. Effectiveness of interventions during NICU hospitalization on the neurodevelopment of preterm infants: a systematic review protocol. Syst Rev. 2017 Nov 3;6(1):225. doi: 10.1186/s13643-017-0613-5. PMID 29100533
- [Background] Malak R, Fechner B, Sikorska D, Rosolek M, Mojs E, Samborski W, Baum E. Application of the Neonatal Behavioral Assessment Scale to Evaluate the Neurobehavior of Preterm Neonates. Brain Sci. 2021 Sep 28;11(10):1285. doi: 10.3390/brainsci11101285. PMID 34679350
- [Background] Aita M, De Clifford Faugere G, Lavallee A, Feeley N, Stremler R, Rioux E, Proulx MH. Effectiveness of interventions on early neurodevelopment of preterm infants: a systematic review and meta-analysis. BMC Pediatr. 2021 Apr 29;21(1):210. doi: 10.1186/s12887-021-02559-6. PMID 33926417
- [Background] Raghupathy MK, Rao BK, Nayak SR, Spittle AJ, Parsekar SS. Effect of family-centered care interventions on motor and neurobehavior development of very preterm infants: a protocol for systematic review. Syst Rev. 2021 Feb 18;10(1):59. doi: 10.1186/s13643-021-01612-w. PMID 33602324